CLINICAL TRIAL: NCT00836927
Title: An Extension Trial of Deforolimus (AP23573; MK-8669), an mTOR Inhibitor, for Patients With Advanced Cancer
Brief Title: Extension Trial of Deforolimus (Ridaforolimus, MK-8669) in Participants With Advanced Cancer (MK-8669-038)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-038; AP23573-08-901 (Other: Ariad Protocol Number); MK-8669-038 (Other: Merck Protocol Number)
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2018-05-03 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Advanced Cancers
MeSH Terms: interventions — ridaforolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ridaforolimus 10 mg Days 1-5 (Experimental): Ridaforolimus 10 mg administered orally once daily on Days 1-5 per week. Participants may continue ridaforolimus intravenous (IV) infusion at the same dose from the parent trial before being switched to ridaforolimus oral tablet.
  Interventions: Drug: Ridaforolimus Tablet; Drug: Ridaforolimus Intravenous (IV) Infusion
- Ridaforolimus 10 mg Days 1-6 (Experimental): Ridaforolimus 10 mg administered orally once daily on Days 1-6 per week. Participants may continue ridaforolimus IV infusion at the same dose from the parent trial before being switched to ridaforolimus oral tablet.
  Interventions: Drug: Ridaforolimus Tablet; Drug: Ridaforolimus Intravenous (IV) Infusion
- Ridaforolimus 20 mg Days 1-5 (Experimental): Ridaforolimus 20 mg administered orally once daily on Days 1-5 per week. Participants may continue ridaforolimus IV infusion at the same dose from the parent trial before being switched to ridaforolimus oral tablet.
  Interventions: Drug: Ridaforolimus Tablet; Drug: Ridaforolimus Intravenous (IV) Infusion
- Ridaforolimus 30 mg Days 1-5 (Experimental): Ridaforolimus 30 mg administered orally once daily on Days 1-5 per week. Participants may continue ridaforolimus IV infusion at the same dose from the parent trial before being switched to ridaforolimus oral tablet.
  Interventions: Drug: Ridaforolimus Tablet; Drug: Ridaforolimus Intravenous (IV) Infusion
- Ridaforolimus 40 mg Days 1-5 (Experimental): Ridaforolimus 40 mg administered orally once daily on Days 1-5 per week. Participants may continue ridaforolimus IV infusion at the same dose from the parent trial before being switched to ridaforolimus oral tablet.
  Interventions: Drug: Ridaforolimus Tablet; Drug: Ridaforolimus Intravenous (IV) Infusion

INTERVENTIONS:
Drug: Ridaforolimus Tablet — Ridaforolimus 10 mg oral tablet
  Other Names: AP23573; MK-8669; ridaforolimus was also known as deforolimus until May 2009
Drug: Ridaforolimus Intravenous (IV) Infusion — Ridaforolimus IV infusion administered once daily for 5 days every 2 weeks in a 28-day cycle (two 2-week courses equals 1 cycle).
  Other Names: AP23573; MK-8669; ridaforolimus was also known as deforolimus until May 2009

SUMMARY:
To describe the long-term safety of deforolimus (ridaforolimus, MK-8669) in participants for whom a clinical benefit has been established in a prior parent trial (MK-8669-013, NCT00060645; MK-8669-016, NCT00112372; and MK-8669-028, NCT00704054) with deforolimus and/or in those who remain in long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Must have participated on a deforolimus (ridaforolimus) parent trial
* Must have derived a clinical benefit from the parent trial
* Is not on any other anti-cancer treatment(s) unless the therapy was allowed on the parent protocol
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 if the participant is scheduled to receive treatment with deforolimus; no requirement if the participant is included for follow-up purposes only
* Participant of childbearing potential must have a negative pregnancy test within 7 days prior to screening and must use approved contraceptive from screening until 30 days after the last dose of study drug
* Signed informed consent

Exclusion Criteria:

* Has not participated on a parent trial
* Women who are to receive study drug who are pregnant or lactating
* Any condition in the Investigator's judgment that renders the participant unable to fully understand and provide informed consent and/or comply with the protocol

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2018-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who continued to receive clinical benefit from ridaforolimus, or who were being followed for long-term safety and efficacy under the following prior protocols were eligible for enrollment into this extension study: MK-8669-013, NCT00060645; MK-8669-016, NCT00112372; and MK-8669-028, NCT00704054.
Pre-assignment Details: Participants may have continued ridaforolimus IV infusion at the same dose from the parent trial before being switched to ridaforolimus oral tablet.
Groups:
- Ridaforolimus 10 mg Days 1-5: Ridaforolimus 10 mg administered orally once daily on Days 1-5 per week.
- Ridaforolimus 10 mg Days 1-6: Ridaforolimus 10 mg administered orally once daily on Days 1-6 per week.
- Ridaforolimus 20 mg Days 1-5: Ridaforolimus 20 mg administered once daily on Days 1-5 per week.
- Ridaforolimus 30 mg Days 1-5: Ridaforolimus 30 mg administered orally once daily on Days 1-5 per week.
- Ridaforolimus 40 mg Days 1-5: Ridaforolimus 40 mg administered orally once daily on Days 1-5 per week.
Period: Overall Study
Arm/Group | Ridaforolimus 10 mg Days 1-5 | Ridaforolimus 10 mg Days 1-6 | Ridaforolimus 20 mg Days 1-5 | Ridaforolimus 30 mg Days 1-5 | Ridaforolimus 40 mg Days 1-5
Started | 3 | 1 | 1 (One participant received ridaforolimus 3 mg IV infusion before being switched to the oral tablet.) | 1 | 1
Completed Dosing Through 03 Apr 2017 | 0 | 1 (Participant continued to receive study drug past the data cut-off date of 03 Apr 2017) | 1 (Participant continued to receive study drug past the data cut-off date of 03 Apr 2017) | 0 | 0
Completed | 0 | 1 (Participant completed treatment by 04 Feb 2018) | 1 (Participant completed treatment by 04 Feb 2018) | 0 | 0
Not Completed | 3 | 0 | 0 | 1 | 1
Not completed — Progressive disease | 2 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ridaforolimus 10 mg Days 1-5 | Ridaforolimus 10 mg Days 1-6 | Ridaforolimus 20 mg Days 1-5 | Ridaforolimus 30 mg Days 1-5 | Ridaforolimus 40 mg Days 1-5 | Total
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 1 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.7 (15.0) | 47.0 | 67.0 | 53.0 | 13.0 | 46.1 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 1 | 6
  Male | 1 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 3 | 1 | 1 | 1 | 0 | 6
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: An adverse event is defined as any unintended or undesirable, noxious, or pathological change, compared to pre-existing conditions, experienced by a participant during a clinical study or the follow-up period, regardless of relationship to study drug. The number of participants who experienced an adverse event is presented.
Time Frame: Up to approximately 2991 days, including 30 days after the last dose (through data cut-off date of 03 Apr 2017)
Population: All participants who received any study drug on this extension protocol according to their actual treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ridaforolimus 10 mg Days 1-5 | Ridaforolimus 10 mg Days 1-6 | Ridaforolimus 20 mg Days 1-5 | Ridaforolimus 30 mg Days 1-5 | Ridaforolimus 40 mg Days 1-5
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 1
Participants | 3 | 1 | 1 | 1 | 1

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD), or death due to any cause, whichever occurred first. Per Response Criteria in Solid Tumors version 1.1 (RECIST 1.1), PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered PD. The PFS for all participants is presented in days.
Time Frame: Up to approximately 2961 days (through data cut-off date of 03 Apr 2017)
Population: All participants who received any study drug on this extension protocol according to their actual treatment.
Measure: Mean (Full Range); unit: Days
Arm/Group | Ridaforolimus 10 mg Days 1-5 | Ridaforolimus 10 mg Days 1-6 | Ridaforolimus 20 mg Days 1-5 | Ridaforolimus 30 mg Days 1-5 | Ridaforolimus 40 mg Days 1-5
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 1
Days | 488.67 [78 to 1297] | 2858 [2858 to 2858] | 2936 [2936 to 2936] | 1142 [1142 to 1142] | 29 [29 to 29]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis will be censored at the date of the last follow-up.
Time Frame: Up to approximately 2991 days (through data cut-off date of 03 Apr 2017)
Population: All participants who received any study drug on this extension protocol according to their actual treatment.
Measure: Mean (Full Range); unit: Days
Arm/Group | Ridaforolimus 10 mg Days 1-5 | Ridaforolimus 10 mg Days 1-6 | Ridaforolimus 20 mg Days 1-5 | Ridaforolimus 30 mg Days 1-5 | Ridaforolimus 40 mg Days 1-5
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 1
Days | 1803.67 [1067 to 2451] | 2933 [2933 to 2933] | 2962 [2962 to 2962] | 2334 [2334 to 2334] | 247 [247 to 247]

4. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: An adverse event is defined as any unintended or undesirable, noxious, or pathological change, compared to pre-existing conditions, experienced by a participant during a clinical study or the follow-up period, regardless of relationship to study drug. The number of participants who discontinued study drug due to an adverse event is presented.
Time Frame: Up to approximately 2961 days (through data cut-off date of 03 Apr 2017)
Population: All participants who received any study drug on this extension protocol according to their actual treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ridaforolimus 10 mg Days 1-5 | Ridaforolimus 10 mg Days 1-6 | Ridaforolimus 20 mg Days 1-5 | Ridaforolimus 30 mg Days 1-5 | Ridaforolimus 40 mg Days 1-5
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrated a confirmed response (Completed Response [CR] or Partial Response [PR]) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment.
Time Frame: Up to approximately 2961 days (through data cut-off date of 03 Apr 2017)
Population: All participants who received any study drug on this extension protocol according to their actual treatment and who experienced a CR or PR.
Measure: Number; unit: Days
Arm/Group | Ridaforolimus 10 mg Days 1-5 | Ridaforolimus 10 mg Days 1-6 | Ridaforolimus 20 mg Days 1-5 | Ridaforolimus 30 mg Days 1-5 | Ridaforolimus 40 mg Days 1-5
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
Days |  |  | 2894 |  |

ADVERSE EVENTS:
Time Frame: Adverse events were collected in the study database for up to approximately 2991 days (including 30 days after the last dose as of data cut-off date 03 Apr 2017). Following closure of the database through 04 Feb 2018 (approximately 307 days), only serious adverse events were collected.
Description: MedDRA preferred terms "Neoplasm Progression", "Malignant Neoplasm Progression" and "Disease Progression" not related to the drug are excluded. All-cause mortality includes deaths not due to an adverse event. Analysis population includes all participants who received any study drug on this extension protocol according to their actual treatment.
Groups:
- Ridaforolimus 10 mg Days 1-5 (Up to Data Cut-Off): Ridaforolimus 10 mg administered orally once daily on Days 1-5 per week.
- Ridaforolimus 10 mg Days 1-6 (Up to Data Cut-Off): Ridaforolimus 10 mg administered orally once daily on Days 1-6 per week.
- Ridaforolimus 20 mg Days 1-5 (Up to Data Cut-Off): Ridaforolimus 20 mg administered once daily on Days 1-5 per week.
- Ridaforolimus 30 mg Days 1-5 (Up to Data Cut-Off): Ridaforolimus 30 mg administered orally once daily on Days 1-5 per week.
- Ridaforolimus 40 mg Days 1-5 (Up to Data Cut-Off): Ridaforolimus 40 mg administered orally once daily on Days 1-5 per week.
- Ridaforolimus 10 mg Days 1-6 (Post Data Cut-Off): Participants remaining on treatment after closure of the study database. Ridaforolimus 10 mg administered orally once daily on Days 1-6 per week.
- Ridaforolimus 20 mg Days 1-5 (Post Data Cut-Off): Participants remaining on treatment after closure of the study database. Ridaforolimus 20 mg administered orally once daily on Days 1-5 per week.
Arm/Group | Ridaforolimus 10 mg Days 1-5 (Up to Data Cut-Off) | Ridaforolimus 10 mg Days 1-6 (Up to Data Cut-Off) | Ridaforolimus 20 mg Days 1-5 (Up to Data Cut-Off) | Ridaforolimus 30 mg Days 1-5 (Up to Data Cut-Off) | Ridaforolimus 40 mg Days 1-5 (Up to Data Cut-Off) | Ridaforolimus 10 mg Days 1-6 (Post Data Cut-Off) | Ridaforolimus 20 mg Days 1-5 (Post Data Cut-Off)
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/1 | 0/1 | 0/1 | 1/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 1/1 | 1/1 | 1/1 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ridaforolimus 10 mg Days 1-5 (Up to Data Cut-Off) (N=3) | Ridaforolimus 10 mg Days 1-6 (Up to Data Cut-Off) (N=1) | Ridaforolimus 20 mg Days 1-5 (Up to Data Cut-Off) (N=1) | Ridaforolimus 30 mg Days 1-5 (Up to Data Cut-Off) (N=1) | Ridaforolimus 40 mg Days 1-5 (Up to Data Cut-Off) (N=1) | Ridaforolimus 10 mg Days 1-6 (Post Data Cut-Off) (N=1) | Ridaforolimus 20 mg Days 1-5 (Post Data Cut-Off) (N=1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ridaforolimus 10 mg Days 1-5 (Up to Data Cut-Off) (N=3) | Ridaforolimus 10 mg Days 1-6 (Up to Data Cut-Off) (N=1) | Ridaforolimus 20 mg Days 1-5 (Up to Data Cut-Off) (N=1) | Ridaforolimus 30 mg Days 1-5 (Up to Data Cut-Off) (N=1) | Ridaforolimus 40 mg Days 1-5 (Up to Data Cut-Off) (N=1) | Ridaforolimus 10 mg Days 1-6 (Post Data Cut-Off) (N=0) | Ridaforolimus 20 mg Days 1-5 (Post Data Cut-Off) (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (14) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Blepharospasm (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | NA | NA
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (3) | 0 (0) | 1 (5) | 0 (0) | NA | NA
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | NA | NA
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (10) | 1 (1) | 1 (1) | 0 (0) | NA | NA
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Fatigue (General disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | NA | NA
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Chest X-ray abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (11) | 1 (3) | 0 (0) | 0 (0) | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | NA | NA
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | NA | NA
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | NA | NA
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All unpublished information that the Sponsor gives to the Investigator shall be kept confidential and shall not be published or disclosed to a third party without the prior written consent of the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-10-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT00836927/Prot_SAP_000.pdf